CLINICAL TRIAL: NCT04250207
Title: A Double-Masked, Randomised, Placebo-Controlled, Parallel-Group, 12 Week, Phase 2 Study to Investigate the Safety and Efficacy of K-321 Eye Drops After Descemetorhexis in Patients With Fuchs Endothelial Corneal Dystrophy
Brief Title: Study to Investigate the Safety and Efficacy of K-321 in Patients With Fuchs Endothelial Corneal Dystrophy (FECD) Following Descemetorhexis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K-321-201
Record Dates: First submitted 2020-01-16; First posted 2020-01-31 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- K-321 QID (Experimental): K-321 Ophthalmic Solution Dose A
  Interventions: Drug: K-321 Solution
- K-321 BID (Experimental): K-321 Ophthalmic Solution Dose B
  Interventions: Drug: K-321 Solution; Drug: Placebo Solution
- Placebo (Placebo Comparator): Vehicle Solution Dose
  Interventions: Drug: Placebo Solution

INTERVENTIONS:
Drug: K-321 Solution — K-321 solution drops
  Arms: K-321 BID; K-321 QID
Drug: Placebo Solution — Placebo solution drops for K-321
  Arms: K-321 BID; Placebo

SUMMARY:
The objective of this study is to investigate the effect of K-321 in patients with Fuchs endothelial corneal dystrophy (FECD) after descemetorhexis.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old at the screening visit (Visit 1).
* Has a diagnosis of FECD at Visit 1.
* Meet all other inclusion criteria outlined in clinical study protocol.

Exclusion Criteria:

* Has a study eye with a history of cataract surgery within 90 days of Visit 1.
* Has a study eye with a history of any previous ocular surgery other than for cataract.
* Meet any other exclusion criteria outlined in clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shona Pendse, MD, MMSc, Study Chair — Kowa Pharma Development Co.
Locations (29):
- United States (19):
  - Jules Stein Eye Institute, Los Angeles, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - UC Davis Eye Center, Sacramento, California
  - Sacramento Eye Consultants, Sacramento, California
  - Gorovoy MD Eye Specialists, Fort Myers, Florida
  - UF Health Eye Center, Gainesville, Florida
  - Chicago Cornea Consultants Ltd, Hoffman Estates, Illinois
  - Arbor Centers For Eyecare, Orland Park, Illinois
  - Price Vision Group, Indianapolis, Indiana
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - W Kellogg Eye Center, Ann Arbor, Michigan
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Eye Associates of New Mexico, Albuquerque, New Mexico
  - NY Langone Health, New York, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Devers Eye Institute, Portland, Oregon
  - Casey Eye Institute - OHSU, Portland, Oregon
  - Vantage EyeCare, LLC, Bala-Cynwyd, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
- Australia (2):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Denmark (2):
  - Rigshospitalet - Glostrup, Glostrup Municipality, Capital
  - Aarhus Universitetshospital, Aarhus
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universität des Saarlandes, Homburg, Saarland
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Instituto Ophthalmologic Fernandez Vega, Oviedo, Principality of Asturias
  - Instituto de Microcirugia Ocular, Barcelona
  - Hospital La Arruzafa, Córdoba

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After obtaining informed consent at Visit 1, the investigator selected one eye as the study eye, and the patient returned for the descemetorhexis operation and random assignment to treatment after 1 to 4 weeks (Visit 2). At Visit 2, eligibility for study participation was confirmed, which included the requirement of a successful descemetorhexis operation which met the inclusion criteria. After eligibility was confirmed, patients were randomly assigned to the 3 treatment groups in a 1:1:1 ratio.
Groups:
- K-321 QID: K-321 ophthalmic solution 4 times daily for 12 Weeks (Morning, Mid-day, Evening, Night).
- K-321 BID: K-321 ophthalmic solution twice daily for 12 Weeks. (Morning: K-321, Mid-day: Placebo, Evening: Placebo, Night: K-321)
- Placebo: Placebo ophthalmic solution four times daily for 12 Weeks. (Morning, Mid-day, Evening, Night)
Period: 12 Week Treatment
Arm/Group | K-321 QID | K-321 BID | Placebo
Started | 21 | 22 | 22
Completed | 21 | 22 | 20
Not Completed | 0 | 0 | 2
Period: 40 Week Follow-up Observation
Arm/Group | K-321 QID | K-321 BID | Placebo
Started | 21 | 22 | 22
Completed | 21 | 21 | 20
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consist of all participants who have a successful descemetorhexis procedure performed, were randomly assigned to receive double-mask study drug, received at least one dose of study drug in the study eye, and have at least one assessment of central corneal ECD performed after the descemetorhexis procedure on the study eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | K-321 QID | K-321 BID | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 22 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (12.28) | 65.1 (9.68) | 65.3 (9.00) | 65.03 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 20 | 49
  Male | 5 | 9 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 2 | 8
  Not Hispanic or Latino | 16 | 21 | 20 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 1 | 1 | 2 | 4
  White | 20 | 19 | 20 | 59
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Central Corneal Endothelial Cell Density (ECD) at Week 12
Description: Change in Central ECD at week 12
Time Frame: Baseline to Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
cells/mm2 | 530.86 (312.453) | 468.02 (322.361) | 228.05 (297.860)
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Test type: Superiority; p = 0.0065, Other (Wilcoxon Rank Sum Test)
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Test type: Superiority; p = 0.0344, Other (Wilcoxon Rank Sum Test)

2. Secondary Outcome: Central Corneal ECD From Baseline to Each Subsequent Visit
Time Frame: Baseline to Week 52
Population: The number of participants analyzed for the outcome measure may differ from the overall number of participants in each group. This discrepancy can be attributed to several factors, including:
  * Missing data: Some participants may have incomplete data due to factors such as missed visits, early withdrawal, or loss to follow-up.
  * Optional visits: Week 2 was an optional visit and saw a smaller number of participants contributing data to specific outcome measures.
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
cells/mm2
  Baseline | 440.01 (774.300) | 319.06 (593.294) | 254.27 (468.027)
  Week 1: number analyzed (Participants) | 20 | 22 | 22
  Week 1 | 0.00 (0.00) | 0.05 (0.218) | 0.05 (0.213)
  Week 2: number analyzed (Participants) | 20 | 22 | 22
  Week 2 | 0.00 (0.00) | 0.05 (0.218) | 0.05 (0.213)
  Week 3 | 131.98 (171.648) | 31.90 (102.749) | 27.49 (127.828)
  Week 5 | 167.36 (176.049) | 167.94 (218.321) | 104.54 (218.264)
  Week 7 | 303.14 (294.919) | 302.95 (232.956) | 79.38 (215.197)
  Week 9 | 370.71 (338.393) | 340.76 (310.264) | 156.04 (278.455)
  Week 12 | 530.86 (312.453) | 468.02 (322.361) | 228.05 (297.860)
  Week 16 | 540.52 (311.004) | 499.77 (358.411) | 286.75 (350.269)
  Week 20 | 655.20 (260.268) | 518.50 (296.094) | 347.21 (313.930)
  Week 24 | 668.22 (313.783) | 541.02 (328.131) | 386.83 (353.840)
  Week 38 | 722.23 (331.954) | 529.65 (303.691) | 391.10 (316.339)
  Week 52 | 751.45 (407.259) | 633.05 (313.372) | 431.79 (327.488)
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Baseline; Test type: Superiority; p = 0.3587, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Baseline; Test type: Superiority; p = 0.5724, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: K-321 QID vs Placebo; Week 1; Test type: Superiority; p = 0.3703, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: K-321 BID vs Placebo; Week 1; Test type: Superiority; p > 0.9999, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: K-321 QID vs Placebo; Week 2; Test type: Superiority; p = 0.3703, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: K-321 BID vs Placebo; Week 2; Test type: Superiority; p > 0.9999, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: K-321 QID vs Placebo; Week 3; Test type: Superiority; p = 0.0257, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: K-321 BID vs Placebo; Test type: Superiority; p = 0.7263, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: K-321 QID vs Placebo; Week 5; Test type: Superiority; p = 0.0607, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: K-321 BID vs Placebo; Week 5; Test type: Superiority; p = 0.0460, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: K-321 QID vs Placebo; Week 7; Test type: Superiority; p = 0.0111, Wilcoxon Rank Sum Test
Statistical Analysis 12: Comparison: K-321 BID vs Placebo; Week 7; Test type: Superiority; p = 0.0011, Wilcoxon Rank Sum Test
Statistical Analysis 13: Comparison: K-321 QID vs Placebo; Week 9; Test type: Superiority; p = 0.0200, Wilcoxon Rank Sum Test
Statistical Analysis 14: Comparison: K-321 BID vs Placebo; Week 9; Test type: Superiority; p = 0.0476, Wilcoxon Rank Sum Test
Statistical Analysis 15: Comparison: K-321 QID vs Placebo; Week 12; Test type: Superiority; p = 0.0065, Wilcoxon Rank Sum Test
Statistical Analysis 16: Comparison: K-321 BID vs Placebo; Week 12; Test type: Superiority; p = 0.0344, Wilcoxon Rank Sum Test
Statistical Analysis 17: Comparison: K-321 QID vs Placebo; Week 16; Test type: Superiority; p = 0.0250, Wilcoxon Rank Sum Test
Statistical Analysis 18: Comparison: K-321 BID vs Placebo; Week 16; Test type: Superiority; p = 0.0733, Wilcoxon Rank Sum Test
Statistical Analysis 19: Comparison: K-321 QID vs Placebo; Week 20; Test type: Superiority; p = 0.0072, Wilcoxon Rank Sum Test
Statistical Analysis 20: Comparison: K-321 BID vs Placebo; Week 20; Test type: Superiority; p = 0.1124, Wilcoxon Rank Sum Test
Statistical Analysis 21: Comparison: K-321 QID vs Placebo; Week 24; Test type: Superiority; p = 0.0199, Wilcoxon Rank Sum Test
Statistical Analysis 22: Comparison: K-321 BID vs Placebo; Week 24; Test type: Superiority; p = 0.2331, Wilcoxon Rank Sum Test
Statistical Analysis 23: Comparison: K-321 QID vs Placebo; Week 38; Test type: Superiority; p = 0.0024, Wilcoxon Rank Sum Test
Statistical Analysis 24: Comparison: K-321 BID vs Placebo; Week 38; Test type: Superiority; p = 0.1672, Wilcoxon Rank Sum Test
Statistical Analysis 25: Comparison: K-321 QID vs Placebo; Week 52; Test type: Superiority; p = 0.0047, Wilcoxon Rank Sum Test
Statistical Analysis 26: Comparison: K-321 BID vs Placebo; Week 52; Test type: Superiority; p = 0.0625, Wilcoxon Rank Sum Test

3. Secondary Outcome: Change From Baseline in Central Corneal Thickness
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
μm
  Week 1: number analyzed (Participants) | 18 | 14 | 18
  Week 1 | 265.57 (125.944) | 250.30 (90.448) | 319.33 (130.570)
  Week 2: number analyzed (Participants) | 19 | 14 | 18
  Week 2 | 237.54 (94.157) | 249.14 (90.636) | 315.18 (131.996)
  Week 3: number analyzed (Participants) | 19 | 18 | 20
  Week 3 | 96.73 (134.360) | 132.63 (152.920) | 201.68 (126.387)
  Week 5: number analyzed (Participants) | 20 | 20 | 21
  Week 5 | 52.71 (109.696) | 32.31 (110.784) | 159.95 (128.295)
  Week 7: number analyzed (Participants) | 20 | 21 | 21
  Week 7 | 42.24 (114.048) | 2.37 (98.340) | 134.83 (132.811)
  Week 9: number analyzed (Participants) | 20 | 21 | 21
  Week 9 | 10.36 (98.235) | -14.23 (60.223) | 116.77 (141.046)
  Week 12: number analyzed (Participants) | 20 | 21 | 21
  Week 12 | 0.59 (86.332) | -22.69 (61.127) | 100.19 (137.191)
  Week 16: number analyzed (Participants) | 20 | 21 | 21
  Week 16 | 2.40 (67.680) | -9.71 (50.918) | 70.00 (132.908)
  Week 20: number analyzed (Participants) | 20 | 21 | 21
  Week 20 | 16.99 (90.440) | -17.70 (46.593) | 70.52 (139.880)
  Week 24: number analyzed (Participants) | 20 | 21 | 21
  Week 24 | 10.60 (78.376) | -27.80 (42.954) | 68.17 (147.116)
  Week 38: number analyzed (Participants) | 20 | 21 | 21
  Week 38 | -12.32 (66.319) | -21.40 (42.525) | 63.09 (149.562)
  Week 52: number analyzed (Participants) | 20 | 21 | 21
  Week 52 | -6.74 (65.888) | -25.88 (44.360) | 55.29 (155.649)
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Week 1; Test type: Superiority; p = 0.2434, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Week 1; Test type: Superiority; p = 0.2126, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: K-321 QID vs Placebo; Week 2; Test type: Superiority; p = 0.0790, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: K-321 BID vs Placebo; Week 2; Test type: Superiority; p = 0.3043, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: K-321 QID vs Placebo; Week 3; Test type: Superiority; p = 0.0357, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: K-321 BID vs Placebo; Week 3; Test type: Superiority; p = 0.0803, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: K-321 QID vs Placebo; Week 5; Test type: Superiority; p = 0.0150, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: K-321 BID vs Placebo; Week 5; Test type: Superiority; p = 0.0012, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: K-321 QID vs Placebo; Week 7; Test type: Superiority; p = 0.0314, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: K-321 BID vs Placebo; Week 7; Test type: Superiority; p = 0.0019, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: K-321 QID vs Placebo; Week 9; Test type: Superiority; p = 0.0170, Wilcoxon Rank Sum Test
Statistical Analysis 12: Comparison: K-321 BID vs Placebo; Week 9; Test type: Superiority; p = 0.0021, Wilcoxon Rank Sum Test
Statistical Analysis 13: Comparison: K-321 QID vs Placebo; Week 12; Test type: Superiority; p = 0.0127, Wilcoxon Rank Sum Test
Statistical Analysis 14: Comparison: K-321 BID vs Placebo; Week 12; Test type: Superiority; p = 0.0014, Wilcoxon Rank Sum Test
Statistical Analysis 15: Comparison: K-321 QID vs Placebo; Week 16; Test type: Superiority; p = 0.0677, Wilcoxon Rank Sum Test
Statistical Analysis 16: Comparison: K-321 BID vs Placebo; Week 16; Test type: Superiority; p = 0.0243, Wilcoxon Rank Sum Test
Statistical Analysis 17: Comparison: K-321 QID vs Placebo; Week 20; Test type: Superiority; p = 0.1867, Wilcoxon Rank Sum Test
Statistical Analysis 18: Comparison: K-321 BID vs Placebo; Week 20; Test type: Superiority; p = 0.0250, Wilcoxon Rank Sum Test
Statistical Analysis 19: Comparison: K-321 QID vs Placebo; Week 24; Test type: Superiority; p = 0.3213, Wilcoxon Rank Sum Test
Statistical Analysis 20: Comparison: K-321 BID vs Placebo; Week 24; Test type: Superiority; p = 0.0298, Wilcoxon Rank Sum Test
Statistical Analysis 21: Comparison: K-321 QID vs Placebo; Week 38; Test type: Superiority; p = 0.1449, Wilcoxon Rank Sum Test
Statistical Analysis 22: Comparison: K-321 BID vs Placebo; Week 38; Test type: Superiority; p = 0.0947, Wilcoxon Rank Sum Test
Statistical Analysis 23: Comparison: K-321 QID vs Placebo; Week 52; Test type: Superiority; p = 0.5181, Wilcoxon Rank Sum Test
Statistical Analysis 24: Comparison: K-321 BID vs Placebo; Week 52; Test type: Superiority; p = 0.1898, Wilcoxon Rank Sum Test

4. Secondary Outcome: Time to Achievement of no Corneal Oedema of Study Eye
Time Frame: Baseline to Week 52
Population: Proportions of patients from the FAS who achieved no corneal edema of the study eye
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Days | 35.0 [22.0 to 64.0] | 51.5 [50.0 to 269.0] | 267.0 [141.0 to 365.0]
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Test type: Superiority; p = 0.0021, Log Rank
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Test type: Superiority; p = 0.1696, Log Rank

5. Secondary Outcome: Proportion of Patients Who Achieved Central Corneal ECD of 700 Cells/mm2 or More at Each Visit
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Participants
  Week 1: number analyzed (Participants) | 20 | 21 | 22
  Week 1 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 3 | 2 | 2
  Week 2 | 0 | 0 | 0
  Week 3: number analyzed (Participants) | 21 | 21 | 20
  Week 3 | 0 | 0 | 0
  Week 5: number analyzed (Participants) | 20 | 22 | 19
  Week 5 | 0 | 0 | 1
  Week 7: number analyzed (Participants) | 20 | 22 | 20
  Week 7 | 3 | 0 | 1
  Week 9: number analyzed (Participants) | 21 | 22 | 18
  Week 9 | 3 | 2 | 2
  Week 12: number analyzed (Participants) | 21 | 21 | 16
  Week 12 | 6 | 4 | 2
  Week 16: number analyzed (Participants) | 21 | 22 | 18
  Week 16 | 6 | 7 | 3
  Week 20: number analyzed (Participants) | 19 | 20 | 12
  Week 20 | 9 | 7 | 3
  Week 24: number analyzed (Participants) | 21 | 18 | 14
  Week 24 | 10 | 8 | 6
  Week 38: number analyzed (Participants) | 18 | 18 | 15
  Week 38 | 12 | 5 | 3
  Week 52: number analyzed (Participants) | 19 | 18 | 15
  Week 52 | 15 | 8 | 5
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Week 5; Test type: Superiority — p-value is based on the Pearson Chi-square test. When the number of responders (Achieved or Not Achieved) is less than 5 in either group, Fisher's exact test is used instead. If Fisher's exact test is used, the unconditional CI for the difference in response rates is provided; p = 0.4872, Chi-square or Fisher exact
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.4634, Chi-square or Fisher exact
Statistical Analysis 3: Comparison: K-321 QID vs Placebo; Week 7; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.6050, Chi-square or Fisher exact
Statistical Analysis 4: Comparison: K-321 BID vs Placebo; Week 7; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.4762, Chi-square or Fisher exact
Statistical Analysis 5: Comparison: K-321 QID vs Placebo; Week 9; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p > 0.9999, Chi-square or Fisher exact
Statistical Analysis 6: Comparison: K-321 BID vs Placebo; Week 9; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p > 0.9999, Chi-square or Fisher exact
Statistical Analysis 7: Comparison: K-321 QID vs Placebo; Week 12; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.4227, Chi-square or Fisher exact
Statistical Analysis 8: Comparison: K-321 BID vs Placebo; Week 12; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.6796, Chi-square or Fisher exact
Statistical Analysis 9: Comparison: K-321 QID vs Placebo; Week 16; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.4642, Chi-square or Fisher exact
Statistical Analysis 10: Comparison: K-321 BID vs Placebo; Week 16; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.4645, Chi-square or Fisher exact
Statistical Analysis 11: Comparison: K-321 QID vs Placebo; Week 20; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.2744, Chi-square or Fisher exact
Statistical Analysis 12: Comparison: K-321 BID vs Placebo; Week 20; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.7026, Chi-square or Fisher exact
Statistical Analysis 13: Comparison: K-321 QID vs Placebo; Week 24; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.7817, Chi-square or Fisher exact
Statistical Analysis 14: Comparison: K-321 BID vs Placebo; Week 24; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.9285, Chi-square or Fisher exact
Statistical Analysis 15: Comparison: K-321 QID vs Placebo; Week 38; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0135, Chi-square or Fisher exact
Statistical Analysis 16: Comparison: K-321 BID vs Placebo; Week 38; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.6992, Chi-square or Fisher exact
Statistical Analysis 17: Comparison: K-321 QID vs Placebo; Week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0135, Chi-square or Fisher exact
Statistical Analysis 18: Comparison: K-321 BID vs Placebo; Week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.5154, Chi-square or Fisher exact

6. Secondary Outcome: Time to Achieve Central Corneal ECD 700 Cells/mm2 or More
Time Frame: Up to 52 Weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Days | 141.0 [83.0 to 363.0] | 181.0 [113.0 to NA] — The curve that represents the upper confidence limits for the failure function lies under 0.50. Therefore, the upper limits of 50th (Median) event time couldn't be estimated. | 273.0 [135.0 to NA] — The curve that represents the upper confidence limits for the failure function lies under 0.50. Therefore, the upper limits of 50th (Median) event time couldn't be estimated.
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Test type: Superiority; p = 0.1209, Log Rank
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Test type: Superiority; p = 0.7116, Log Rank

7. Secondary Outcome: Number of Patients Who Achieved Corneal Thickness Less Than or Equal to Baseline Corneal Thickness
Time Frame: Baseline up to 52 Weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Participants
  Week 1: number analyzed (Participants) | 18 | 14 | 18
  Week 1 | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 3 | 1 | 1
  Week 2 | 0 | 0 | 0
  Week 3: number analyzed (Participants) | 19 | 18 | 20
  Week 3 | 5 | 3 | 1
  Week 5: number analyzed (Participants) | 20 | 20 | 20
  Week 5 | 8 | 9 | 2
  Week 7: number analyzed (Participants) | 20 | 21 | 20
  Week 7 | 11 | 13 | 3
  Week 9: number analyzed (Participants) | 20 | 21 | 19
  Week 9 | 11 | 16 | 5
  Week 12: number analyzed (Participants) | 20 | 21 | 18
  Week 12 | 13 | 17 | 5
  Week 16: number analyzed (Participants) | 20 | 21 | 17
  Week 16 | 14 | 13 | 6
  Week 20: number analyzed (Participants) | 20 | 20 | 14
  Week 20 | 12 | 14 | 8
  Week 24: number analyzed (Participants) | 20 | 20 | 16
  Week 24 | 13 | 17 | 9
  Week 38: number analyzed (Participants) | 18 | 19 | 16
  Week 38 | 15 | 16 | 10
  Week 52: number analyzed (Participants) | 18 | 18 | 16
  Week 52 | 14 | 15 | 13
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0915, Chi-square or Fisher exact
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.3282, Chi-square or Fisher exact
Statistical Analysis 3: Comparison: K-321 QID vs Placebo; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0648, Chi-square or Fisher exact
Statistical Analysis 4: Comparison: K-321 BID vs Placebo; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0310, Chi-square or Fisher exact
Statistical Analysis 5: Comparison: K-321 QID vs Placebo; Week 7; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0187, Chi-square or Fisher exact
Statistical Analysis 6: Comparison: K-321 BID vs Placebo; Week 7; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0036, Chi-square or Fisher exact
Statistical Analysis 7: Comparison: K-321 QID vs Placebo; Week 9; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0687, Chi-square or Fisher exact
Statistical Analysis 8: Comparison: K-321 BID vs Placebo; Week 9; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0016, Chi-square or Fisher exact
Statistical Analysis 9: Comparison: K-321 QID vs Placebo; Week 12; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0218, Chi-square or Fisher exact
Statistical Analysis 10: Comparison: K-321 BID vs Placebo; Week 12; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0013, Chi-square or Fisher exact
Statistical Analysis 11: Comparison: K-321 QID vs Placebo; Week 16; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0348, Chi-square or Fisher exact
Statistical Analysis 12: Comparison: K-321 BID vs Placebo; Week 16; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.1028, Chi-square or Fisher exact
Statistical Analysis 13: Comparison: K-321 QID vs Placebo; Week 20; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.8677, Chi-square or Fisher exact
Statistical Analysis 14: Comparison: K-321 BID vs Placebo; Week 20; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.4401, Chi-square or Fisher exact
Statistical Analysis 15: Comparison: K-321 QID vs Placebo; Week 24; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.5926, Chi-square or Fisher exact
Statistical Analysis 16: Comparison: K-321 BID vs Placebo; Week 24; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0732, Chi-square or Fisher exact
Statistical Analysis 17: Comparison: K-321 QID vs Placebo; Week 38; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.2497, Chi-square or Fisher exact
Statistical Analysis 18: Comparison: K-321 BID vs Placebo; Week 38; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.2453, Chi-square or Fisher exact
Statistical Analysis 19: Comparison: K-321 QID vs Placebo; Week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p > 0.9999, Chi-square or Fisher exact
Statistical Analysis 20: Comparison: K-321 BID vs Placebo; Week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p > 0.9999, Chi-square or Fisher exact

8. Secondary Outcome: Proportion of Patients Who Achieve No Corneal Oedema of Study Eye by Visit
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Participants
  Week 1 | 0 | 0 | 0
  Week 2 | 0 | 0 | 0
  Week 3 | 8 | 0 | 1
  Week 5 | 11 | 4 | 1
  Week 7 | 11 | 12 | 2
  Week 9 | 14 | 12 | 2
  Week 12 | 17 | 12 | 2
  Week 16 | 16 | 13 | 2
  Week 20 | 15 | 12 | 7
  Week 24 | 17 | 13 | 8
  Week 38 | 17 | 13 | 10
  Week 52 | 17 | 13 | 13
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0093, Chi-square or Fisher exact
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Week 3; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p > 0.9999, Chi-square or Fisher exact
Statistical Analysis 3: Comparison: K-321 QID vs Placebo; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0006, Chi-square or Fisher exact
Statistical Analysis 4: Comparison: K-321 BID vs Placebo; Week 5; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.3449, Chi-square or Fisher exact
Statistical Analysis 5: Comparison: K-321 QID vs Placebo; Week 7; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0028, Chi-square or Fisher exact
Statistical Analysis 6: Comparison: K-321 BID vs Placebo; Week 7; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0028, Chi-square or Fisher exact
Statistical Analysis 7: Comparison: K-321 QID vs Placebo; Week 9; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0001, Chi-square or Fisher exact
Statistical Analysis 8: Comparison: K-321 BID vs Placebo; Week 9; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0028, Chi-square or Fisher exact
Statistical Analysis 9: Comparison: K-321 QID vs Placebo; Week 12; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, Chi-square or Fisher exact
Statistical Analysis 10: Comparison: K-321 BID vs Placebo; Week 12; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0028, Chi-square or Fisher exact
Statistical Analysis 11: Comparison: K-321 QID vs Placebo; Week 16; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, Chi-square or Fisher exact
Statistical Analysis 12: Comparison: K-321 BID vs Placebo; Week 16; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0011, Chi-square or Fisher exact
Statistical Analysis 13: Comparison: K-321 QID vs Placebo; Week 20; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0094, Chi-square or Fisher exact
Statistical Analysis 14: Comparison: K-321 BID vs Placebo; Week 20; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.1281, Chi-square or Fisher exact
Statistical Analysis 15: Comparison: K-321 QID vs Placebo; Week 24; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0051, Chi-square or Fisher exact
Statistical Analysis 16: Comparison: K-321 BID vs Placebo; Week 24; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.1313, Chi-square or Fisher exact
Statistical Analysis 17: Comparison: K-321 QID vs Placebo; Week 38; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0268, Chi-square or Fisher exact
Statistical Analysis 18: Comparison: K-321 BID vs Placebo; Week 38; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.3652, Chi-square or Fisher exact
Statistical Analysis 19: Comparison: K-321 QID vs Placebo; Week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.1854, Chi-square or Fisher exact
Statistical Analysis 20: Comparison: K-321 BID vs Placebo; Week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p > 0.9999, Chi-square or Fisher exact

9. Secondary Outcome: Time to Return of Corneal Thickness to Less Than or Equal to Baseline Cornea Thickness
Time Frame: Baseline up to Week 52
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Days | 50 [35.0 to 110.0] | 50.0 [34.0 to 66.0] | 165.0 [112.0 to 366.0]
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Test type: Superiority; p = 0.0259, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Test type: Superiority; p = 0.0068, Wilcoxon Rank Sum Test

10. Secondary Outcome: Percent Change of Central Corneal Thickness From Baseline to Each Subsequent Visit
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | K-321 QID | K-321 BID | Placebo
Number analyzed (Participants) | 21 | 22 | 22
Percent
  Week 1: number analyzed (Participants) | 18 | 14 | 18
  Week 1 | 45.76 (23.191) | 41.48 (15.582) | 51.41 (21.687)
  Week 2: number analyzed (Participants) | 3 | 1 | 1
  Week 2 | 39.03 (10.916) | 36.77 (NA) — Number of Participant Analyzed is one in each Arm. Therefore SD can't be estimated. | 40.97 (NA) — Number of Participant Analyzed is one in each Arm. Therefore SD can't be estimated.
  Week 3: number analyzed (Participants) | 19 | 18 | 20
  Week 3 | 16.50 (22.581) | 21.85 (25.600) | 32.39 (20.422)
  Week 5: number analyzed (Participants) | 20 | 20 | 20
  Week 5 | 9.24 (19.101) | 5.31 (17.421) | 25.67 (21.873)
  Week 7: number analyzed (Participants) | 20 | 21 | 20
  Week 7 | 7.58 (19.744) | 0.43 (15.276) | 20.84 (22.228)
  Week 9: number analyzed (Participants) | 20 | 21 | 19
  Week 9 | 2.51 (18.451) | -2.28 (9.442) | 14.55 (18.954)
  Week 12: number analyzed (Participants) | 20 | 21 | 17
  Week 12 | 0.73 (15.895) | -3.65 (9.467) | 10.70 (17.611)
  Week 16: number analyzed (Participants) | 20 | 21 | 16
  Week 16 | 0.74 (11.936) | -1.65 (7.955) | 2.91 (11.967)
  Week 20: number analyzed (Participants) | 19 | 20 | 14
  Week 20 | 3.85 (17.227) | -3.64 (6.726) | 1.93 (14.291)
  Week 24: number analyzed (Participants) | 20 | 20 | 15
  Week 24 | 2.27 (14.662) | -5.42 (5.927) | 2.79 (16.807)
  Week 38: number analyzed (Participants) | 18 | 19 | 15
  Week 38 | -3.63 (7.992) | -4.98 (5.229) | -2.00 (9.969)
  Week 52: number analyzed (Participants) | 18 | 18 | 15
  Week 52 | -2.90 (8.634) | -5.63 (5.614) | -3.68 (11.182)
Statistical Analysis 1: Comparison: K-321 QID vs Placebo; Week 1; Test type: Superiority; p = 0.4435, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: K-321 BID vs Placebo; Week 1; Test type: Superiority; p = 0.3402, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: K-321 QID vs K-321 BID; Week 2; Test type: Superiority; p > 0.9999, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: K-321 QID vs Placebo; Week 3; Test type: Superiority; p = 0.0655, Wilcoxon Rank Sum Test
Statistical Analysis 5: Comparison: K-321 BID vs Placebo; Week 3; Test type: Superiority; p = 0.0903, Wilcoxon Rank Sum Test
Statistical Analysis 6: Comparison: K-321 QID vs Placebo; Week 5; Test type: Superiority; p = 0.0216, Wilcoxon Rank Sum Test
Statistical Analysis 7: Comparison: K-321 BID vs Placebo; Week 5; Test type: Superiority; p = 0.0020, Wilcoxon Rank Sum Test
Statistical Analysis 8: Comparison: K-321 QID vs Placebo; Week 7; Test type: Superiority; p = 0.0676, Wilcoxon Rank Sum Test
Statistical Analysis 9: Comparison: K-321 BID vs Placebo; Week 7; Test type: Superiority; p = 0.0029, Wilcoxon Rank Sum Test
Statistical Analysis 10: Comparison: K-321 QID vs Placebo; Week 9; Test type: Superiority; p = 0.0335, Wilcoxon Rank Sum Test
Statistical Analysis 11: Comparison: K-321 BID vs Placebo; Week 9; Test type: Superiority; p = 0.0053, Wilcoxon Rank Sum Test
Statistical Analysis 12: Comparison: K-321 QID vs K-321 BID; Week 12; Test type: Superiority; p = 0.0608, Wilcoxon Rank Sum Test
Statistical Analysis 13: Comparison: K-321 BID vs Placebo; Week 12; Test type: Superiority; p = 0.0071, Wilcoxon Rank Sum Test
Statistical Analysis 14: Comparison: K-321 QID vs Placebo; Week 16; Test type: Superiority; p = 0.4406, Wilcoxon Rank Sum Test
Statistical Analysis 15: Comparison: K-321 BID vs Placebo; Week 16; Test type: Superiority; p = 0.1716, Wilcoxon Rank Sum Test
Statistical Analysis 16: Comparison: K-321 QID vs Placebo; Week 20; Test type: Superiority; p = 0.9856, Wilcoxon Rank Sum Test
Statistical Analysis 17: Comparison: K-321 BID vs Placebo; Week 20; Test type: Superiority; p = 0.2229, Wilcoxon Rank Sum Test
Statistical Analysis 18: Comparison: K-321 QID vs K-321 BID; Week 24; Test type: Superiority; p = 0.8817, Wilcoxon Rank Sum Test
Statistical Analysis 19: Comparison: K-321 BID vs Placebo; Test type: Superiority; p = 0.2081, Wilcoxon Rank Sum Test
Statistical Analysis 20: Comparison: K-321 QID vs Placebo; Week 38; Test type: Superiority; p = 0.7335, Wilcoxon Rank Sum Test
Statistical Analysis 21: Comparison: K-321 BID vs Placebo; Week 38; Test type: Superiority; p = 0.5367, Wilcoxon Rank Sum Test
Statistical Analysis 22: Comparison: K-321 QID vs K-321 BID; Week 52; Test type: Superiority; p = 0.5550, Wilcoxon Rank Sum Test
Statistical Analysis 23: Comparison: K-321 BID vs Placebo; Week 52; Test type: Superiority; p = 0.8718, Wilcoxon Rank Sum Test

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Treatment emergent adverse events (TEAE) were any adverse event that occurred or worsened after the first dose of study treatment.
Arm/Group | K-321 QID | K-321 BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/22 | 3/22
Other Adverse Events (participants affected / at risk) | 12/21 | 11/22 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | K-321 QID (N=21) | K-321 BID (N=22) | Placebo (N=22)
Appendicitis (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Terminal ileitis (Gastrointestinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alcohol rehabilitation (Surgical and medical procedures) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-321 QID (N=21) | K-321 BID (N=22) | Placebo (N=22)
Conjunctival hyperaemia (Eye disorders) | 3 | 3 | 0
Corneal oedema (Eye disorders) | 4 | 2 | 7
Eye pruritus (Eye disorders) | 1 | 3 | 0
Vision blurred (Eye disorders) | 1 | 2 | 3
Photophobia (Eye disorders) | 1 | 2 | 2
Corneal disorder (Eye disorders) | 0 | 2 | 1
Eye irritation (Eye disorders) | 0 | 2 | 1
Foreign body sensation in eyes (Eye disorders) | 0 | 2 | 1
Diplopia (Eye disorders) | 0 | 2 | 0
Eye pain (Eye disorders) | 0 | 2 | 5
Visual acuity reduced (Eye disorders) | 1 | 3 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Eye allergy (study eye) (Eye disorders) | 2 | 0 | 0
Corneal degeneration (Eye disorders) | 2 | 1 | 1
Eye allergy (non-study eye) (Eye disorders) | 2 | 0 | 0
Punctate keratitis (Eye disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must review proposed publication 60 days before submission. Sponsor can request revisions and delay publication for up to 60 days to file patents. Sponsor may also require removal of specific information (other than study results).

DOCUMENTS (5):
  • Study Protocol: Ver. 1.0 (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT04250207/Prot_000.pdf
  • Study Protocol: Ver. 2.0 (2019-12-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT04250207/Prot_001.pdf
  • Statistical Analysis Plan: Ver. 1.0 (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04250207/SAP_002.pdf
  • Statistical Analysis Plan: Ver. 2.0 (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04250207/SAP_003.pdf
  • Statistical Analysis Plan: Ver. 2.0 Addendum (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04250207/SAP_004.pdf